CLINICAL TRIAL: NCT03742843
Title: A Multi-omics Study on the Tumorigenesis of Adenomyosis
Brief Title: A Multi-omics Study of Adenomyosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: AM-OMICS
Record Dates: First submitted 2018-11-09; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Adenomyosis; Endometriosis; Ectopic Endometrium; Eutopic Endometrium; Genomics; Transcriptomics; Metabolomics
MeSH Terms: conditions — Adenomyosis; Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An 8 ml peripheral venous blood, and 50 μL adenomyosis/endometriosis tissue and tissue adjacent to adenomyosis/endometriosis will be collected from eligible patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group of adenomyosis: Patients with adenomyosis with or without endometriosis
  Interventions: Combination Product: A multi-omics analysis
- Group of endometriosis: Patients with endometriosis without adenomyosis
  Interventions: Combination Product: A multi-omics analysis
- Group of control: Patients without adenomyosis or endometriosis
  Interventions: Combination Product: A multi-omics analysis

INTERVENTIONS:
Combination Product: A multi-omics analysis — A multi-omics analysis including whole exome sequencing, transcriptomics and metabolomics for eutopic and ectopic endometrium

SUMMARY:
This study aims to analyze the multi-omics results between eutopic endometrium, adenomyosis and endometriosis of patients diagnosed of adenomyosis with and without endometriosis. The multi-omics profiles include whole exome sequencing, analysis of transcriptomics and metabolomics. A comprehensive multi-omics will reveal the pathogenesis of adenomyosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed adenomyosis and/or endometriosis
* Signed an approved informed consents
* Feasible for biopsy

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with adenomyosis and/or endomtriosis and feasible for biopsy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2020-11-23 (Estimated); Study Completion 2020-11-23 (Estimated)

PRIMARY OUTCOMES:
Frequencies of somatic driving mutations | Two years
  The differences of distributions and frequencies of somatic driving mutations will be compared between eutopic endometrium and ectopic endometrium by whole exome sequencing.

SECONDARY OUTCOMES:
Frequencies of alteration of RNA expression | Two years
  The alteration of RNA expression, including mRNA, miRNA, and lncRNA, will be compared between eutopic endometrium and ectopic endometrium by transcriptome sequencing.
Frequencies of alteration of protein expression and signal pathway | Two years
  The alteration of protein expression and signal pathway will be compared between eutopic endometrium and ectopic endometrium by metabolomic sequencing
Progression-free survival | Five years
  Progression-free survival between patients with differential expressed multi-omics will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China